CLINICAL TRIAL: NCT03634449
Title: Comparing the Gastroesophageal Reflux on Endotracheal Intubation or the I-gel- Second Generation Supraglottic Airway Device in the Pneumoperitoneum and Trendelenburg Surgical Setting
Brief Title: Risks of Gastroesophageal Reflux in the Endotracheal Intubation or the I-gel
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 201806063RINB
Record Dates: First submitted 2018-08-09; First posted 2018-08-16 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2018-08

CONDITIONS: Gastroesophageal Reflux in Laparoscopy

STUDY DESIGN:
Intervention Model Description: one group using the endotracheal tube one group using the i-gel
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- i-gel (Experimental): After anesthetic durg given, i-gel, a supraglottic airway devices with a gastric suction channel, will be inserted into the patients' airway.
  Interventions: Device: i-gel
- endotracheal tube (Active Comparator): After anesthetic durg given, the endotracheal tube, traditional use for protect airway during the laparoscopic surgery, will be inserted into the patients' airway.
  Interventions: Device: endotracheal tube

INTERVENTIONS:
Device: i-gel — i-gel is a supraglottic airway devices with a gastric suction channel.
  Arms: i-gel
Device: endotracheal tube — Endotracheal intubation is a traditional use for protect airway during the laparoscopic surgery.
  Arms: endotracheal tube

SUMMARY:
In the use of the second supraglottic airway device- i-gel in the laparoscopic pneumoperitoneum and Trendelenburg (LPT) surgical positioning, our data reported that the leak fraction in the i-gel group was higher than in the endotracheal tube group.1 These air leak may be gone into the GI tract and cause the gastric distension resulting in the increasing risk of aspiration. Few studies investigated whether the risk of occurrence of the gastroesophageal reflux (GER), the changes of the lower esophageal sphincter (LES) while the GER occurred, and the stomach fullness in the i-gel group than in the endotracheal tube group.

We aim to observe the changes of gastroesophageal function parameters by esophageal manometry, pH impedance, and intra-abdominal pressure before and after laparoscopic pneumoperitoneum during anesthesia, all via the second SADs.

DETAILED DESCRIPTION:
Background: In the use of the second supraglottic airway device- i-gel in the laparoscopic pneumoperitoneum and Trendelenburg (LPT) surgical positioning, our data reported that the leak fraction in the i-gel group was higher than in the endotracheal tube group.1 These air leak may be gone into the GI tract and cause the gastric distension resulting in the increasing risk of aspiration. Few studies investigated whether the risk of occurrence of the gastroesophageal reflux (GER), the changes of the lower esophageal sphincter (LES) while the GER occurred, and the stomach fullness in the i-gel group than in the endotracheal tube group. The LES is the important physiological mechanisms that prevent regurgitation and aspiration. The previous study has been investigated that LES would have adaptive response in using the endotracheal tube in the LPT setting. However, the change of LES pressure and gastroesophageal reflux during the LPT surgical settings using the i-gel is still unknown.

The esophageal manometry has pressure sensor to measure the LES pressure. The combined esophageal multichannel intraluminal impedance and pH monitoring (MII -pH) could not only detect the acidic reflux or weakly acidic reflux, but also the height of the regurgitant. We also used the abdominal echo in check the gastric volume before and after the surgery.

Objectives: we aimed to compare the changes of lower esophageal sphincter pressure (LESP) and the occurrence of the GER during the LPT setting by esophageal manometry and MII-pH monitor between the endotracheal tube (ETT) and the i-gel group. The gastric volume before and after surgery has been checked by abdominal echo. We also observed the respiratory parameters changes while the GER occurred.

Patients and methods: Consecutive patients who will receive scheduled laparoscopic surgery under general anesthesia and aged from 20 to 80 years old will be enrolled. All subjects provide basic demographic data. The patients have been randomized into the i-gel or ETT group by sealing envelope. After induction, the MII-pH monitor has been pre-attached to the esophageal manometry. Then they will be inserted into the esophagus. The patients have received the ETT or i-gel. Then the respiratory parameters were collected by the GE S/5 Compact Anesthesia Monitor (GE Healthcare, Helsinki, Finland) with a spirometry tube (GE Healthcare, Helsinki, Finland) and D-lite sensor (GE Healthcare, Helsinki, Finland). The data have been continuous recorded. There were four time point of the LESP measured: (1)T1, after induction (without muscle relaxant) (2)T2, ETT or i-gel intubation (3)T3, after LPT setting (4) T4, off LPT setting.

Expected result: We will compared the difference between the patients receiving the i-gel or ETT group about the (1) the changes of LESP in the above four time point (2) the occurrence of the GER and the relationship between the LES and GER (3) gastric volume before and after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will receive scheduled surgery with laparoscopic pneumoperitoneum and Trendelenburg (LPT) setting under general anesthesia
* Aged from 20-80 years old

Exclusion Criteria:

* Major systemic disease, such as congestive heart failure, liver cirrhosis, end stage renal disease and malignancy.
* Patients who have the risk of difficult ventilation or intubation.
* pregnant women
* coagulopathy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-08-13 (Actual); Primary Completion 2019-10-13 (Estimated); Study Completion 2020-09-13 (Estimated)

PRIMARY OUTCOMES:
gastroesophageal reflux occurence | during the surgery
  occurence of the gastroesophageal reflux

SECONDARY OUTCOMES:
lower esophageal sphincter change | during the surgery
  lower esophageal sphincter change during the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Chih-Jun Lai, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
due to the privacy of the individual participant data of our patients, we cannot share their data to other researchers.
  The raw data will be kept very carefully in our research team.